CLINICAL TRIAL: NCT05714475
Title: Multicentre Retrospective Study on Pancreas Resection for Colorectal Cancer Metastasis
Brief Title: Pancreas Resection for Colorectal Metastasis: Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Francesco Palmieri, MD, Principal investigator, Ospedale Generale Di Zona Moriggia-Pelascini
Other Study IDs: MP1
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pancreas Metastases; Colorectal Cancer
Keywords: pancreas; pancreatectomy; pancreas resection; colorectal metastasis; whipple; adenocarcinoma; follow up
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreas resection for colorectal metastasis: Patient underwent a pancreas resection (whipple, distal pancreasectomy ...) with inclusion criteria. Criteria
  Inclusion Criteria:
  * Isolated pancreatic metastases from Colorectal cancer
  * Previous surgery for colorectal cancer
  * Surgically manageable lesions: duodenal-pancreatectomy surgical removal of metastatic repetitions in pancreas
  * Other procedures:
  total-pancreatectomy distal-pancreatectomy other metastases resection
  * R0 resection
  * no signs of peritoneal metastasis or tumor manifestations outside of the pancreas.
  * CT Scan before surgery
  Exclusion Criteria:
  * metastases from different malignancies
  * other malignancies
  * surgically unmanageable lesions
  * Multiple synchronous colorectal metastasis
  Interventions: Procedure: Pancreas surgery

INTERVENTIONS:
Procedure: Pancreas surgery — Criteria
  Inclusion Criteria:
  * Isolated pancreatic metastases from Colorectal cancer
  * Previous surgery for colorectal cancer
  * Surgically manageable lesions: duodenal-pancreatectomy surgical removal of metastatic repetitions in pancreas
  pancreaticoduodenectomy total-pancreatectomy distal-pancreatectomy other metastases resection

SUMMARY:
The aim of this study is to collect data from different centres to obtain a larger case series and enable a better definition of the outcomes after pancreatic metastasectomy from primary colorectal cancer. To evaluate the possible benefits of surgery, we intend to retrospectively analyze the outcome of patients in whom pancreatic metastases have been surgically treated.

Primary objective;

1. To evaluate feasibility and safety of pancreas resection in metastatic colorectal cancer
2. To evaluate oncological outcome at six months from surgical procedure

Secondary objective:

1. To evaluate oncological outcome at 12 months from surgical procedure

DETAILED DESCRIPTION:
Metastases to the Pancreas are quite rare and account for less than 5% of pancreatic malignancies diagnosed in living patients.

In autopsy cases of malignant tumours, the incidence of pancreatic secondary tumours reaches 15%.

The metastases are predominantly of epithelial origin, most commonly from lung, stomach, small bowel, colon-rectum, kidney , breast , liver , ovary ,melanoma and urinary bladder.

It is largely described that resection of isolated metastasis to the lung or liver from primary tumour leads to improved survival; yet there is no consensus about the benefit of pancreas resection for metastases and the gold standard treatment is still not well defined.

The lack of data for pancreas metastases resections depends on low incidence and high perioperative risks. However, the improvement in morbidity and mortality rates after pancreaticoduodenectomy made the indication for this operation acceptable.

One of the larger series concluded that an aggressive surgical approach might be warranted if the patient can be rendered free of disease.

The majority of case series referred to renal cell carcinoma and resection for CCR are episodic. However there are several reports of solitary resected pancreatic metastases from colorectal cancer There is currently very limited experience with the surgical resection of isolated pancreatic colorectal metastases, and the role of surgery in the management of these patients is still debated.

To date, no prospective randomized or case-controlled studies have been performed to evaluate the role of surgical resection. Additionally, many of the existing retrospective studies are limited because of the small number of patients who were treated during prolonged periods of time.

Aim of the study The aim of this study is to collect data from different centres to obtain a larger case series and enable a better definition of the outcomes after pancreatic metastasectomy from primary colorectal cancer. To evaluate the possible benefits of surgery, the investigators intend to retrospectively analyze the outcome of patients in whom pancreatic metastases have been surgically treated.

The investigators launched the study aiming at demonstrating that pancreatic resection for colorectal metastases may be a safe and feasible procedure in selected patients and may provide long-term survival. The investigators sought to address the role of surgical resection and survival benefit from surgery. The investigators suppose to achieve a good prognosis with a median survival close to that observed after resection of hepatic metastases.

The guidelines for the treatment of colorectal cancer recommend resection of hematogenous metastases if they are deemed resectable.

Study design This study is an international multicenter retrospective cohort study to assess the outcomes of patients that underwent pancreas resection for solitary colorectal metastasis.

Aim of surgical interventions is to remove metastases in association to radical lymphadenectomy thus to achieve R0 result.

Patient data will be retrospectively analyzed and demographic characteristics, comorbidity status, clinical and radiological findings, treatment strategies , 30-day morbidity and mortality, oncological outcomes at 6 and 12 months will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Isolated pancreatic metastases from Colorectal cancer
* Previous surgery for colorectal cancer
* Surgically manageable lesions: duodenal-pancreatectomy surgical removal of metastatic repetitions in pancreas
* Other procedures:

total-pancreatectomy distal-pancreatectomy other metastases resection

* R0 resection
* no signs of peritoneal metastasis or tumor manifestations outside of the pancreas.
* CT Scan before surgery

Exclusion Criteria:

* metastases from different malignancies
* other malignancies
* surgically unmanageable lesions
* Multiple synchronous colorectal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent pancreas surgery for colorectal metastasis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  assessed by the number of patients with pancreas resection deceased within 30-days from the surgical intervention
30-day morbidity | 30 days
  assessed by the number of patients with pancreatic resection who experienced any type of postoperative complication within 30-days from the surgical intervention
Overall survival | 6 months
  6 moths survival 3. Survival : 6 moths survival 4. Disease free survival at 6 months
Disease free survival | 6 months
  disease free survival at 6 months

SECONDARY OUTCOMES:
Overall survival (12) | 12 months
  Overall survival at 12 months
Disease free survival (12) | 12 months
  disease free survival at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di zona Moriggia Pelascini, Gravedona, Como, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR